CLINICAL TRIAL: NCT04246515
Title: The Effect of Blood Flow Restriction Training on the Mechanical Properties of Hamstring Injuries: A Prospective, Randomised Clinical Trial Using Supersonic Shear Wave Elastography
Brief Title: The Effect of Blood Flow Restriction Training on Hamstring Elasticity After Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B670201940629
Record Dates: First submitted 2020-01-21; First posted 2020-01-29 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Hamstring Injury
Keywords: Hamstring injury; Shear Wave Elastography; Blood Flow Restriction
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blood Flow Restriction Training (Experimental): As from week 2 in the rehabilitation proces, this experimental group will receive exercises in combination with blood flow restriction. While occluding the vascular flow of the limb (startpoint = above the injury site), participants will perform 3 exercises: wall squat, leg press and bridge (3 sets of 30 repetitions). These blood flow restricted exercises are always on top of the classic rehabilitation.
  Interventions: Device: Blood Flow Restriction Training
- Sham Blood Flow Restriction Training (Sham Comparator): The same description as the experimental arm is applicable here. However, The Blood Flow restriction material will be attached to the injured limb without occluding the vascular blood flow.
  Interventions: Device: Sham Blood Flow Restriction Training
- Classic rehabilitation (Active Comparator): This group will undergo the classic rehabilitation program.
  Interventions: Other: Classic rehabilitation

INTERVENTIONS:
Device: Blood Flow Restriction Training — Vascular occlusion of the injured limb.
  Other Names: Vascular occlusion Training
  Arms: Blood Flow Restriction Training
Device: Sham Blood Flow Restriction Training — Blood Flow Restriction material will be attached to the limb without vascular occlusion.
  Arms: Sham Blood Flow Restriction Training
Other: Classic rehabilitation — Classic rehabilitation protocol after a hamstring injury consisiting out of stretching, strength, core stability,...
  Arms: Classic rehabilitation

SUMMARY:
The aim of this study is to investigate the effect of Blood Flow Restriction Training on the elasticity of the hamstring muscle after an acute injury. Therefore a group of football players with a recent hamstring strain injury (HSI) will be recruited and randomly assigned in one of the three following groups:

Experimental group: Classic rehabilitation + Blood Flow Restriction Training

Sham group: Classic rehabilitation + sham Blood Flow Restriction Training

Control group: Classic rehabilitation

The study procedure will be as followed:

1. HSI (onset) -> recruitment via football clubs, physiotherapy practices, leaflets,…
2. MRI scan (day 0-4) -> injury location, grade and extend (The British Athletics Medical Team Classification)
3. Shear Wave Elastography (SWE) measurement (day 0-4) of the injured site and the exact same location at the contralateral leg.
4. Rehabilitation in one of the three groups + Testing

   At the first therapy session a standardized initial assessment sheet will be filled in comprising of all the necessary information regarding patient information and history (recent hamstring injury and past injuries) . Furthermore, a weekly assessment of the strongest predictors of rehabilitation duration will be conducted. Between day 12 and 16 a second shear wave elastographic measurement will be performed.
5. Return to play (RTP)

   The RTP decision will be made by the head physician and the attending physiotherapist. The decision will be based on clearly predefined criteria. At moment of RTP a third shear wave elastographic measurement will be performed.
6. Follow-up

The football players will be contacted regularly by phone to inquire about possible re-injuries, this for a period of 6 months after injury onset. At week 12 after injury onset, a fourth and last shear wave elastographic measurement will be performed.

The evolution of the hamstring elasticity and other outcome measures will be compared between groups and also within groups between the injured leg and the healthy contralateral leg.

DETAILED DESCRIPTION:
In this study, 90 participants with an acute hamstring strain injury will participate. Age restrictions will be delimited between 18 and 35 years old to rule out age-related confounding factors. Potential participants will be excluded from this study if they had a history of hamstring injuries, or a recent severe trauma or surgery in the lower extremity. A hamstring injury is defined as a football-related injury in the posterior thigh muscle region, preventing a player from participating in training or competition for at least 1 week. In addition, any contra-indication for occluding vascular flow (such as hypertension, risk factors for and/or history of cardiovascular pathologies or thromboembolism, surgery, fractures, severe obesity,…) will entail an immediate exclusion from the study.

Within 4 days after the onset of a suspected HSI the participant will undergo a magnetic resonance (MR) scan in order to acquire more insight in the severity, location and extend of the injury. The British Athletics Medical Team Classification will be used to classify HSI on the basis of grade (1: small tear, 2: moderate tear, 3: extensive tear or 4: complete tear) and injury site (a: myofascial, b: MTJ or c: tendon). [Pollock et al.2014] Each participant will be assigned an unique number and subsequently randomly assigned to either the control, experimental treatment or sham group by using an online research randomizer (http://www.randomizer.org) which is already used in previous literature [van der Horst et al. 2015]. This will result in a total of 30 participants per treatment group. The experimental group will perform, on top of a classic rehabilitation protocol, exercises while occluding the vascular blood flow. The use of low-intensity exercises with vascular blood flow restriction (BFR) has been found, in previous studies, to induce the same hypertrophic muscle adaptations as high-intensity exercises without BFR. The combination of increased metabolic stress, due to an Ischemic and hypoxic muscular environment, and exercise induced mechanical tension is suggested to be responsible for this effect. [Hughes et al. 2017] The patients in the sham BFR group will receive the same protocol as the experimental group with the exception of not inflating the Blood flow restriction cuff, causing no real vascular occlusion. Furthermore, the intervention in the control group will consist out of a classic rehabilitation program suitable for treating a hamstring injury. Shortly after the MR scan, still in the first week after injury onset, a shear wave elastography measurement of the injured site and at exact same location at non-injured site will be performed. Appendicular to the first, three more elastographic measurements will be performed at fixed moments in time: between day 12 and 16, at moment of return to play (RTP) and at week 12 after injury onset. All the participants will undergo a standardized rehabilitation protocol in one of the three groups until the medical team cleared the patient for returning to sport participation, based on clearly defined and standardised criteria. Tests and questionnaires for evaluation of hamstring strength, flexibility, pain and functionality will be conducted at three major moments in the rehabilitation process: within the first therapy session, weekly during the complete rehabilitation process and at moment of return to play. After RTP, athletes will be contacted regularly, until six months after injury onset, to determine the number of re-injuries. A questionnaire concerning demographic and anthropometric data, sport activities and injury history will be completed by the participants, prior to the testing protocol, as these factors will be additionally investigated for their possible influence on the primary outcome measures. The aim of the study is to investigate the effect of vascular occlusion (Blood Flow Restriction Training), within the rehabilitation program, on the healing proces (outcome measures predictive for the duration of the rehabilitation: average pain at each therapy session, eccentric mid and outer range strength, total painful palpation length, maximal hip flexion active knee extension test) and especially on the elasticity of the injured hamstring muscle tissue (measured with shear wave elastography).

ELIGIBILITY:
Inclusion Criteria:

* Acute hamstring strain injury
* Male
* Adult (18+) between 18 and 35 years old

Exclusion Criteria:

* History of hamstring injuries
* Recent severe trauma or surgery in the lower extremity
* Any contra-indication for occluding vascular flow (such as hypertension, risk factors for and/or history of cardiovascular pathologies or thromboembolism, surgery, fractures, severe obesity,…)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only men will be included as this gender population is the most susceptible for the development of hamstring injuries.
Enrollment: 90 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of elasticity | From date of randomization until 12 weeks.
  Change of the Shear Modulus of the injured site of the hamstring from onset untill 12 weeks.
Time to return to play | From injury onset until moment of return to play, up to an average of 3 weeks.
  Time between injury onset and moment of return to play. Return to play is the moment when the athlete is cleared for sport participation by the medical staff based on 4 standardized criteria: 1. No pain on palpation 2. Pain free full Range of Motion (ROM) 3. Max (ecc) strength difference 10 % 4. Symptom-free completion of rehab program and repeated maximal (30m) sprinting.

SECONDARY OUTCOMES:
Pain on palpation and average pain at each therapy session | Weekly from fist therapy session until moment of return to play, up to an average of 3 weeks.
  Pain Visual Analogue Scale (VAS). The pain VAS is a unidimensional measure of pain intensity with the use of a Likert scale from 0 to 10, with 0 = no pain and 10 = worst possible pain.
Eccentric strength | Weekly from fist therapy session until moment of return to play, up to an average of 3 weeks.
  Eccentric strength of the injured hamstring muscle
Flexibility | Weekly from fist therapy session until moment of return to play, up to an average of 3 weeks.
  Flexibility of the injured hamstring muscle using the Maximal Hip Flexion Active Knee Extension Test (MHFAKE)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Witvrouw, Prof. dr., Principal Investigator — Department of Rehabilitation Sciences, Ghent University
Locations (1):
- Department of rehabilitation sciences, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No